CLINICAL TRIAL: NCT00183339
Title: A Randomized, Placebo-controlled Trial of Fluoxetine in Preschool Children
Brief Title: Early Intervention With Fluoxetine in Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U54MH066418 (NIH); U54MH066418 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-16 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Autistic Disorder
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo, liquid solution flexible dose 0.5 to 5ml every morning (AM)
  Interventions: Drug: Placebo
- fluoxetine (Experimental): Fluoxetine, 20mg/5ml solution, flexible dose 0.5 to 5ml every AM
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Between 2 mg per day and 20 mg per day of liquid fluoxetine will be given in the morning using a flexible dosing strategy, following a 36-week dose titration schedule.
  Other Names: Prozac
  Arms: fluoxetine
Drug: Placebo — Between 0.5ml per day and 5ml per day of liquid placebo will be given in the morning using a flexible dosing strategy, following a 36-week dose titration schedule.
  Arms: Placebo

SUMMARY:
This study is a pilot study to evaluate the feasibility and safety of conducting a year long, double-blind, placebo-controlled trial of fluoxetine in pre-school children to enhance developmental processes in core areas impacted by autism.

DETAILED DESCRIPTION:
Autism, a brain disorder that affects a small percentage of Americans, often results in a lifetime of impaired thinking, feeling, and social functioning. The disorder generally becomes apparent in children by the age of 3. Autism typically affects a person's ability to communicate, form relationships with others, and respond appropriately to the external world. Some people with autism can function at a relatively high level, with speech and intelligence intact. Others have serious cognitive impairments and language delays, and some never speak. This study will assess the safety and effectiveness of treating autistic children with fluoxetine to enhance developmental processes in core areas impacted by autism.

Each participant was randomly assigned to treatment with double-blinded placebo or fluoxetine for 12 months. After initial screening and randomization, participants were assessed every two weeks for approximately the first 3 months, or until the dose of medication is stabilized. After this initial period, they were assessed on a monthly basis. Dosing was flexible as determined by the adverse and beneficial responses to treatment although there was a suggested titration schedule.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism

Exclusion Criteria:

* Diagnosis of Asperger Syndrome, Rett Syndrome, Childhood Disintegrative Disorder, or Pervasive Development Disorder-Not Otherwise Specified
* Informed that treatment with a selective serotonin reuptake inhibitor (SSRI) is medically inadvisable
* Need for ongoing psychotropic medication (except for diphenhydramine, clonidine, or melatonin for sleep)
* Recent use of stimulants within 5 days prior to enrollment
* Ongoing need for or recent use of most psychotropic medications within 14 days of enrollment
* Recent initiation of specialized educational, behavioral, or diet intervention for autism in the month prior to enrollment

Ages: 30 Months to 58 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants who received placebo solution between .5ml and 5.0ml
- Fluoxetine: Participants who received liquid fluoxetine 2-20 mg (of 4mg/1ml solution) in AM using a flexible dose strategy and planned 36 week titration schedule
Period: Overall Study
Arm/Group | Placebo | Fluoxetine
Started | 10 | 8
Completed | 4 | 4
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants will take the placebo
- Fluoxetine: Participants will take liquid fluoxetine 2-20 mg
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluoxetine | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 8 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 44.0 (6.6) | 42.6 (8.1) | 43.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recruitment
Description: In order for a larger trial with similar design to be feasible a number of factors needed to be examined. The first was whether families would enroll very young children with ASD into a year long blinded medication study. To determine this we examined the average number of months to randomize 1 participant per site. We calculated this (as total # months required for recruitment* 2sites ) /[ # participants randomized ] and compared it to the typical # of months required to recruit an older child with ASD for a double-blind 12 week placebo controlled medication study, which is typically about 1.2 months at each of the sites involved in the study.
Time Frame: 19 months
Measure: Number; unit: months/participant at 1 site
Arm/Group | Placebo | Fluoxetine
Number analyzed (Participants) | 10 | 8
months/participant at 1 site | 2.1 | 2.1

2. Secondary Outcome: Rate of Attrition
Description: The percentage of participants who discontinued treatment prior to completion of the 12 month study
Time Frame: Measured at Month 12
Measure: Number; unit: percent of group that discontinued early
Groups:
- Placebo: participants who were treated with flexible dose placebo solution
- Fluoxetine: Participants treated with flexible dose fluoxetine solution
Arm/Group | Placebo | Fluoxetine
Number analyzed (Participants) | 10 | 8
percent of group that discontinued early | 60 | 50

3. Secondary Outcome: Change From Baseline to 12 Months in Total Score on Caregiver Strain Questionnaire
Description: This is a caregiver completed measure that assesses the extent to which the caregiver feels care of the participant influences the caregiver's and other family members' emotional states and/or activities. There are a total of 22 items rated from 1 - not at all to 5 - very much (with one item reverse scored). Total score is the sum of all the items (with one item reverse scored). There are three subscales objective strain -12 items, internalized subjective strain 6 items, externalized subjective 4 items. The total score can range from a minimum of 0 - no strain at all, to 110 all items rated as very much.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluoxetine: participants who were treated with flexible dose (2-20mg/D) fluoxetine solution
Arm/Group | Placebo | Fluoxetine
Number analyzed (Participants) | 10 | 8
units on a scale | 0.8 (2.5) | -1.86 (2.3)

4. Secondary Outcome: Change From Baseline to Month 12 in Aberrant Behavior Checklist Irritability Subscale Score (ABC-I)
Description: The Aberrant Behavior Checklist (ABC) is a caregiver completed rating scale that assesses problem behaviors frequently seen in individuals with developmental disabilities. There are a total of 58 items on 5 subscales that are rated from 0 - not at all a problem to 3 - problem is severe in degree. The ABC-I consists of 15 items that reflect mood swings, self-injury and aggression. The subscale score is the sum of the score on each of the 15 items. The minimum score on the ABC-I is 0 and the maximum score is 45. Higher scores reflect more severe behavioral problems. A score > or = to 18 is generally considered clinically significant.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fluoxetine
Number analyzed (Participants) | 10 | 8
units on a scale | -0.70 (2.9) | -8.50 (10.6)

ADVERSE EVENTS:
Time Frame: 12 months (The course of treatment for each participant in the trial)
Groups:
- Fluoxetine: participants who were treated with flexible dose fluoxetine solution, 2-20mg per day
Arm/Group | Placebo | Fluoxetine
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 9/10 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Fluoxetine (N=8)
Severe Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Fluoxetine (N=8)
Nosebleed (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cold/Flu/other systemic infection (Infections and infestations) | 7 (7) | 6 (6)
Earache (Ear and labyrinth disorders) | 3 (3) | 3 (3)
other eye disorders (Eye disorders) | 0 (0) | 3 (3)
gastroenteritis (Gastrointestinal disorders) | 6 (6) | 6 (6)
allergies (Immune system disorders) | 3 (3) | 4 (4)
intentional injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Local Infection (Infections and infestations) | 1 (1) | 0 (0)
weight increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
aggression (Psychiatric disorders) | 4 (4) | 5 (5)
Other infection (Infections and infestations) | 2 (2) | 1 (1)
enuresis (Renal and urinary disorders) | 2 (2) | 5 (5)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Sensory Sensitivity (General disorders) | 1 (1) | 1 (1)
Sexual (General disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
insomnia (General disorders) | 5 (5) | 5 (5)
irritability (Nervous system disorders) | 4 (4) | 3 (3)
mood lability (Psychiatric disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
It took twice as long to recruit subjects for a study in children 30-58 months than it generally takes to recruit older children. It is possible to maintain subjects in double-blind trails for extended periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No